CLINICAL TRIAL: NCT05638451
Title: Phase 2 Study to Evaluate the Efficacy and Safety of Sintilimab in Combination With Bevacizumab and Temozolomide in Recurrent Glioblastoma (GBM) Patients
Brief Title: Sintilimab in Combination With Bevacizumab and Temozolomide in Recurrent Glioblastoma (GBM) Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Junde Zhang
Record Dates: First submitted 2022-11-27; First posted 2022-12-06 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2023-06

CONDITIONS: Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — sintilimab; Bevacizumab; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintilimab and Bevacizumab and Temozolomide (Experimental): single arm study
  Interventions: Drug: Sintilimab plus Bevacizumab and Temozolomide

INTERVENTIONS:
Drug: Sintilimab plus Bevacizumab and Temozolomide — 200mg Sintilimab plus 10mg/kg Bevacizumab very 3 weeks 200 mg/m2/day Temozolomide on days 1-5 out of a 28 days schedule

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Sintilimab in combination with Bevacizumab and Temozolomide in subjects with recurrent glioblastoma.

DETAILED DESCRIPTION:
This is a phase 2,open-label, multicenter, single-arm study designed to evaluate the efficacy and safety of Sintilimab in combination with Bevacizumab and Temozolomide in subjects with recurrent glioblastoma.

A total of 30 patients will be enrolled in the study and administered Sintilimab in combination with Bevacizumab and Temozolomide. The study treatment will be continued for up to 4 cycles and Sintilimab was maintained until a progression of disease or unacceptable toxicity is confirmed.

ELIGIBILITY:
Inclusion Criteria:

1. Molecular pathological diagnosis was high-grade glioma (2016 World Health Organization (WHO） Grade Ⅲ or Ⅳ);
2. Age 18 - 70 years old, Karnofsky performance status （KPS） score ≥ 70, and the expected survival period is more than 3 months;
3. Primary supratentorial glioblastoma with first or second recurrence
4. Imaging confirmed recurrence (according to RANO criteria);
5. The time of the first medication after enrollment should be more than 4 weeks away from the surgery or the last radiotherapy;
6. Confirmed progression time is ≥4 weeks from the last drug treatment (including adjuvant temozolomide chemotherapy after the completion of concurrent chemoradiotherapy);
7. If the patient is on hormone therapy, the hormone dose must be stable or reduced for at least 7 days before the baseline MRI examination;
8. Major organ function within 7 days prior to treatment, meeting the following criteria:

(1) Routine blood test standards (without blood transfusion within 14 days):

1. Hemoglobin (HB) ≥90 g/L;
2. Absolute neutrophil count (ANC) ≥ 1.5×10^9/L;
3. Platelet (PLT) ≥ 90×10^9/L; (2) Biochemical examination shall meet the following standards:
4. Total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN);
5. Alanine aminotransferase (ALT) and aspartate aminotransferase AST ≤ 2.5 ULN, if with liver metastasis, ALT and AST ≤ 5ULN;
6. Serum creatinine (Cr) ≤1.5 ULN and creatinine clearance rate (CCr) ≥ 60 ml/min; (3) Echocardiography: Left ventricular ejection fraction (LVEF) ≥ lower limit of normal (50%); (4) International normalized ratio (INR), partial thromboplastin time (APTT), prothrombin time (PT) ≤1.5 ULN; 9. Patients voluntarily joined the study and signed informed consent.

Exclusion Criteria:

1. Prior treatment with immunotherapy;
2. Patients who have had or are currently suffering from other malignant tumors or solid organ or bone marrow transplantation within 5 years. Excludes cured cervical carcinoma in situ, non-melanoma skin cancer, and superficial bladder tumors;
3. Baseline MRI indicates the risk of cerebral hemorrhage or hernia in the past or recent;
4. Pulmonary embolism or deep vein thrombosis within 2 months
5. Unstable angina pectoris, myocardial infarction within past 12 months. Grade 2 or greater congestive heart failure
6. Peptic ulcer, abdominal fistula, gastrointestinal perforation, or abdominal abscess within past 6 months
7. Patients with any physical signs or history of bleeding, regardless of severity;
8. Uncontrollable high blood pressure
9. Patients with liver cirrhosis, decompensated liver disease, active hepatitis or chronic hepatitis;
10. Renal failure requires hemodialysis or peritoneal dialysis;
11. Known history of active infectious pneumonia and active tuberculosis.
12. Requiring escalating or chronic supraphysiologic doses of corticosteroids (> 4 mg dexamethasone daily) for control of disease
13. Allergic reaction to bevacizumab or any of its excipients
14. Diagnosis of immunodeficiency, including human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)
15. Active autoimmune disease requiring systemic treatment (i.e., disease modifiers, corticosteroids, or immunosuppressive drugs) within past 2 years. Replacement therapy (such as thyroxine, insulin, or physiologic corticosteroid replacement for adrenal or pituitary insufficiency, etc.) is not considered a systemic form of therapy.
16. Pregnancy or breastfeeding, or pregnancy or birth during the expected test period, from the pre-screening or screening visit until 120 days after the last dose of test treatment.
17. Unable to undergo brain MRI (i.e., pacemaker or any other MRI contraindications).
18. According to the judgment of the investigator, there are concomitant diseases that seriously endanger the patient's safety or affect the patient's completion of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival rate at 6 months | Up to two years
  Progression free survival by iRANO criteria

SECONDARY OUTCOMES:
Progression free survival | Up to two years
  the time interval from entry to tumor progression, Progression free survival (PFS) by iRANO criteria
Overall survival | Up to two years
  the time interval from entry to death from any cause
Objective response rate | Up to two years
  rate of Complete Response +Partial Response
Disease control rate | Up to two years
  rate of Complete Response +Partial Response+Stable Disease
Median duration of Karnofsky Performance Status(KPS) ≥ 70 | Up to two years
  Median duration of KPS ≥ 70 during progression-free survival
Frequency and severity of treatment-related adverse events | Up to two years
  Frequency and severity of treatment-related adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Median duration of stable/improved quality of life assessed by EORTC QLQ-C30 | Up to two years
  the time interval from entry to change of ≥10 points on the EORTC QLQ-C30 without further improvement or disease progression or death
Absolute counts and ratios of immune cell subtypes | Day 1 and Day 29 of each cycle
  Changes of absolute counts and ratios of immune cell subtypes

CONTACTS AND LOCATIONS:
Overall Officials: Junde Zhang, MD, Principal Investigator — Zhujiang Hospital
Locations (1):
- southern medical university affiliated Zhujiang Hospital, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No